CLINICAL TRIAL: NCT04238117
Title: Laser Acupuncture Therapy in Postpartum Low Back Pain: A Prospective Randomized Controlled Study
Brief Title: Laser Acupuncture Therapy in Postpartum Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8G0941
Record Dates: First submitted 2020-01-14; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Lower Back Pain; Postpartum Period
Keywords: Laser acupuncture therapy; Low back pain; Postpartum; low-level laser therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LA group (Experimental): The participants in LAT group underwent 10 sessions of LAT over 2 weeks, using a gallium aluminum arsenide Laser Pen. The participants in the LAT group received 0.375 J of energy at each of the following acupoints bilaterally: BL23 (Shenshu, B2), BL25 (Dachangshu, B2), BL26 (Guanyuanshu, B2), BL40 (Weizhong, B2) and SP6 (Sanyinjiao, B2).
  Interventions: Procedure: Laser acupuncture treatment
- Control group (No Intervention): The participants of the control group received standard obstetric care.

INTERVENTIONS:
Procedure: Laser acupuncture treatment — Laser acupuncture therapy (LAT) is a noninvasive technique that involves stimulation of traditional acupoints with low intensity, non thermal laser irradiation.
  Arms: LA group

SUMMARY:
Over half of women after giving birth have low back pain (LBP), however, LBP is often accepted as a normal part of postpartum. Unsolved low back pain undoubtedly affects women's physical health and may be negatively affect their psychological health. This study was aimed to investigate the efficacy of laser acupuncture therapy (LAT) in postpartum LBP. Postpartum women with LBP admitted at a postpartum care center were recruited and randomly assigned to the intervention group or the control group. The participants in the intervention group underwent 10 sessions/2 weeks of LAT and received standard obstetric care. The participants in the control group only received standard obstetric care. Primary outcome measurements were Visual Analogue Scale (VAS) for pain and salivary cortisol values. Secondary outcome measurements were Chinese versions of the Roland and Morris Disability Questionnaire (RMDQ), Oswestry Disability Index (ODI) version 2.1and the Perceived Stress Scale (PSS).

ELIGIBILITY:
Inclusion Criteria:

1. Age not less than 20 years
2. Women postpartum within one month
3. Low back pain with visual analogue scale (VAS) score ≧1
4. Low back pain was not relieved by rest for 30 minutes.

Exclusion Criteria:

1. with systemic diseases
2. with cancers
3. with psychiatric diseases
4. under treatment for severe pain by a physician.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale (VAS) for pain | 2 weeks
  record VAS score for pain before intervention and 2 weeks after intervention
Change in salivary cortisol values | 2 weeks
  record Salivary cortisol values before intervention and 2 weeks after intervention

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire (RMDQ) | 2 weeks
  The RMDQ is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.
Chinese version of Oswestry Disability Index (ODI) | 2 weeks
  The ODI includes 1 item on pain and 9 items on physical activity of daily living (personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). The total scores ranged from 0 to 40, higher scores indicated greater limitation of physical activities.
Perceived stress (PSS) | 2 weeks
  PSS containes 7 items with positive subscales and 7 items with negative subscales. Each item is rated from 0 to 4 (0 = never, 4 = very often).

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ting Liu, Principal Investigator — Department of Chinese Medicine, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No